CLINICAL TRIAL: NCT05869578
Title: Registry of Patients Subjected to the Perioperative Care of the Anesthesia Service of Clinica Alemana of Santiago Chile
Brief Title: Registry of Anesthesia and Perioperative Medicine
Acronym: RAMP
Status: Not yet recruiting | Type: Observational
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Sponsor
Other Study IDs: UIEC1166
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Complication; Perioperative/Postoperative Complications; Anesthesia Morbidity; Anesthesia; Adverse Effect; Anesthesia Complication; Anesthesia; Reaction
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anesthesia Intervention — Patients exposed to any anesthesia intervention will be assessed to whether the exposure to anesthesia confers a risk for perioperative outcomes

SUMMARY:
To assess mortality and morbidity associated to anesthesia interventions

DETAILED DESCRIPTION:
Currently evidence-based medicine is one of the most important tools guiding our medical practice. Part of this evidence has been generated from clinical records, which has allowed access to large databases from which relevant information has been obtained for perioperative risk stratification, searching for complications, having specific information on procedures, among others.

A clear example, especially useful daily in anesthesia work, is the NSQIP score, a tool that allows calculating perioperative risk according to the conditions of the patient and the surgery. NSQIP score is considered to make decisions in both the American and the European guidelines for preoperative evaluation for surgery.

Latin-American or Chilean databases are not available at the present time. Chile lacks of population perioperative databases, methodology and practice of medicine outcomes records, thus making necessary the generation of a retrospective/prospective registry.

The investigators expect that this registry will allow the collection of perioperative information appropriate to characterize the Chilean population, observe its evolution, and detect risk factors. Moreover, this registry will grant the investigators the means to design new research studies that may allow them to gather medical evidence of superior quality, thus benefiting patients with the best and safest interventions and procedures.

ELIGIBILITY:
Inclusion Criteria:

* All individuals
* Individuals agreeing to participate in the study by signing a consent

Exclusion Criteria:

* The subjects who had insufficient data in their files

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of all ages being admitted at Clinica Alemana de Santiago that will require or were in care by an anesthesiologist.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2035-01-01 (Estimated); Study Completion 2045-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate in the postoperative period | 30 days
  Posoperative mortality of individuals exposed to any anesthesia related intervention or event
All-cause mortality rate in the posoperative period | one year
  Posoperative mortality of individuals exposed to any anesthesia related intervention or event
Number of patients presenting a complication in the posoperative period | 30 days
  Perioperative morbidity of individuals exposed to any anesthesia related intervention or event.
Number of patients who needed rehospitalization in the posoperative period | 7 days after primary discharge
  Posoperative rehospitalization rate of individuals exposed to any anesthesia related intervention or event, after primary discharge
Number of deaths in the postoperative period after readmission | up to 30 days
  In-hospital mortality of patients that were readmitted after primary discharge

SECONDARY OUTCOMES:
Change from baseline in pain, as measured by the visual analog scale (VAS) | Baseline pre-intervention VAS, postoperative/intervention 1 hour VAS, postoperative/intervention 24 hour VAS
  Scores are measured on a 10-point VAS. The VAS ranges from 0 to 10 with 0 indicating no pain, and higher scores indicating greater pain.
Number of patients that develops postoperative acute kidney injury, as measured by Kidney Disease Improving Global Outcomes (KIDGO)-2012 serum creatinine criteria | 7 and 30 days
  Criteria for developing acute kidney injury are:
  Increase in serum creatinin by ≽0.3 mg/dl (≽26.5lmol/l) within 48hours; or Increase in serum creatinine ≽1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or Urine volume < 0.5ml/kg/h for 6hours.
Number of patients that develops postoperative Major Acute Cardiac Events (MACE), as defined by the American Heart Association | 7 and 30 days
  Criteria for MACE are the development of any of the following conditions Non-fatal stroke Non-fatal myocardial infarction Cardiovascular death
Number of patients that develop posoperative chronic pain as measured by visual analog scale | 3, 6, and 12 months
  Scores are measured on a 10-point VAS. The VAS ranges from 0 to 10 with 0 indicating no pain, and higher scores indicating greater pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Abdel-Kader AK, Eisenkraft JB, Katz DJ. Overview and Limitations of Database Research in Anesthesiology: A Narrative Review. Anesth Analg. 2021 Apr 1;132(4):1012-1022. doi: 10.1213/ANE.0000000000005346. PMID 33346984
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, De Hert S, Ford I, Gonzalez Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luescher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Uva MS, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur J Anaesthesiol. 2014 Oct;31(10):517-73. doi: 10.1097/EJA.0000000000000150. No abstract available. PMID 25127426
- [Background] Gupta PK, Gupta H, Sundaram A, Kaushik M, Fang X, Miller WJ, Esterbrooks DJ, Hunter CB, Pipinos II, Johanning JM, Lynch TG, Forse RA, Mohiuddin SM, Mooss AN. Development and validation of a risk calculator for prediction of cardiac risk after surgery. Circulation. 2011 Jul 26;124(4):381-7. doi: 10.1161/CIRCULATIONAHA.110.015701. Epub 2011 Jul 5. PMID 21730309
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 9;130(24):2215-45. doi: 10.1161/CIR.0000000000000105. Epub 2014 Aug 1. No abstract available. PMID 25085962
- [Background] Bosco E, Hsueh L, McConeghy KW, Gravenstein S, Saade E. Major adverse cardiovascular event definitions used in observational analysis of administrative databases: a systematic review. BMC Med Res Methodol. 2021 Nov 6;21(1):241. doi: 10.1186/s12874-021-01440-5. PMID 34742250